CLINICAL TRIAL: NCT05930405
Title: Comparative Analysis of Programmed Intermittent Epidural Bolus Versus Continuous Epidural Infusion on Postoperative Recovery Quality Following Video-Assisted Thoracoscopic Surgery: A Multicenter, Prospective, Double-Blind, Randomised Controlled Trial
Brief Title: Effect of the PIEB Versus CEI on the Quality of Postoperative Recovery in Patients Undergoing VATS Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, RenChun Lai, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-FXY-062
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Video-assisted Thoracic Surgery
Keywords: Programmed intermittent epidural bolus; Continuous epidural infusion; QoR-15; Epidural anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- programmed intermittent epidural bolus group (Experimental): All subjects received a standardised epidural solution containing 0.2% ropivacaine and 0.4（male）/0.3（famale）μg/ml sufentanil with or without PCEA (4 mL). The PIEB group is programmed for intermittent infusion with （0.1*kg）ml pumped every two hours. The lockout time for both groups is 60 min.
  Interventions: Procedure: programmed intermittent epidural bolus
- continuous epidural infusion group (Active Comparator): All subjects received a standardised epidural solution containing 0.2% ropivacaine and 0.4（male）/0.3（famale）μg/ml sufentanil with or without PCEA (4 mL). The CEI group was infused continuously at a rate of （0.05*kg）ml/h. The lockout time for both groups was 60 min.
  Interventions: Procedure: continuous epidural infusion

INTERVENTIONS:
Procedure: programmed intermittent epidural bolus — Bolus a certain amount of liquid at fixed intervals according to a predetermined procedure
  Other Names: PIEB
  Arms: programmed intermittent epidural bolus group
Procedure: continuous epidural infusion — continuous epidural infusion
  Other Names: CEI
  Arms: continuous epidural infusion group

SUMMARY:
In recent years, lobectomy under VATS(Video-assisted thoracic surgery,VATS) has gradually emerged, but there is still a proportion of patients with postoperative pain that affects their postoperative recovery. Epidural analgesia (EA) , the gold standard for postoperative analgesia in thoracic surgery, is currently administered in two ways: 1) continuous epidural infusion 2) programmed intermittent epidural bolus. The former is currently the commonly used method of anesthetic infusion, while the latter has been better studied in obstetrics and major abdominal surgery, but is still unclear in thoracic medicine. This paper aims to investigate the impact of both drug delivery methods on the quality of postoperative recovery in patients undergoing lobectomy by VATS.

DETAILED DESCRIPTION:
In recent years, video-assisted thoracic surgery (VATS) has largely matured and gained widespread acceptance. Patients undergoing VATS have been reported to have less postoperative pain and a better quality of life. VATS has fewer overall post-operative complications, shorter hospital stays and lower rates of blood transfusion than conventional open surgery. However, about 38% of patients who underwent VATS were still reported to have severe postoperative pain. The placement of a thoracic drain increases the level of post-operative pain, especially when the patient breathes deeply, moves around or coughs, making the patient afraid to cooperate with deep breathing or coughing after surgery, thus increasing the chance of post-operative atelectasis and lung infection.

Epidural analgesia (EA) is the 'gold standard' for postoperative analgesia in the thoracic surgery and is an important component of multimodal analgesia in thoracic surgery. Continuous epidural infusion (CEI) of local anesthetic combined with patient-controlled analgesia (PCA) is an effective method of post-operative analgesia in thoracic surgery. However, CEI has some disadvantages, such as increased consumption of local anesthetic and limited distribution area of anesthetic, which does not suppress pain during deep breathing or coughing in the postoperative period very well, resulting in poor appetite and reduced quality of recovery. Programmed intermittent epidural bolus (PIEB) is an epidural analgesia modality that has emerged in recent years and has been more comprehensively studied in the field of postoperative analgesia in obstetrics. PIEB mode has been shown to provide better analgesia and lower consumption of local anesthetic compared to the traditional CEI mode.

The current study of PIEB in thoracic surgery under VATS is still unclear and we wanted to investigate the effect of procedural intermittent epidural bolus (PIEB) versus continuous epidural infusion (CEI) on the quality of recovery in patients undergoing lobectomy by VATS. The trial was divided into two groups, with the control group (CEI group) using a continuous epidural infusion and the trial group (PIEB group) using a programmed intermittent epidural infusion. All subjects received a standardised epidural solution containing 0.2% ropivacaine and 0.4（male）/0.3（famale）μg/ml sufentanil. The CEI group was infused continuously at a rate of 0.05*kg ml/h, while the PIEB group was programmed for intermittent infusion with 0.1*kg pumped every two hours. The PCEA is 4ml in both groups. The lockout time for both groups was 60 min. The maximum infusion dosage of the both groups is 10ml/h. Heart rate, ECG, pulse oximetry, invasive blood pressure, and end-expiratory carbon dioxide partial pressure (ETCO2) are routinely monitored on admission. Prior to induction of anaesthesia, ultrasound-assisted epidural puncture placement in the mid-thoracic segment (T5/6 or T6/7 or T7/8) is performed and the success of placement is judged using the disappearance of resistance method. The epidural catheter was placed 5 cm cephalad and 3 mL of 1.5% lidocaine was injected epidurally as a test dose to rule out inadvertent vessel entry and dural breach. This was followed by an epidural push of 10-20 mL of 0.2% ropivacaine with a test plane in the T1-T10 range. General anesthesia was induced with intravenous dexmedetomidine (0.5 ug/kg), propofol (2 mg/kg), sufentanil (0.2 ug/kg) and cis-atracurium (0.15 mg/kg). Anesthesia is maintained with 4ug/ml propofol in TCI model, with additional cis-atracurium as required, followed by additional epidural 0.2 % ropivacaine at the discretion of the anesthetist and recorded as appropriate. Vasoactive drugs may be used as appropriate to maintain blood pressure fluctuations within ±20% of basal blood pressure. The QoR15 rating scale (Quality of Recovery-15, QoR15) is one of the main methods currently used to evaluate postoperative recovery and is a valid, reliable and responsive patient-centred prognostic indicator that is highly acceptable to both patients and clinicians. Therefore, we used the 24h postoperative QoR15 score as the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Proposed lobectomy under VATS under general anesthesia with tracheal intubation
2. Agree to use epidural analgesia after surgery
3. ASA Ⅰ- Ⅲ grade
4. BMI 18.5-30 kg/m2
5. Age 18-65 years old

Exclusion Criteria:

1. Preoperative refusal of surgery due to accident or subjective
2. Neurological dysfunction
3. contraindications to intralesional anesthesia
4. history of preoperative opioid use
5. Patients with abnormal preoperative pain and pain score (NRS) > 3
6. Patients taking sedative hypnosis, anti-anxiety, and antidepressant drugs for a long time before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
QoR15 score at 24 hours after surgery | Day 1 after surgery
  QoR15 score at 24 hours after surgery

SECONDARY OUTCOMES:
QoR15 score rating at 24, 48 and 72 hours after surgery | 3 days after surgery
  QoR15 score rating at 24, 48 and 72 hours after surgery
QoR15 score at 48 and 72 hours after surgery | second and third days after surgery
  QoR15 score at 48 and 72 hours after surgery
NRS scores at rest or during coughing at 24, 48 and 72 hours after surgery | 3 days after surgery
  NRS scores at rest or during coughing at 24, 48 and 72 hours after surgery
Number of nighttime PCEA at 24, 48 and 72 hours after surgery | 3 days after surgery
  Number of nighttime PCEA at 24, 48 and 72 hours after surgery
Total number of PCEAs at 24, 48 and 72 hours after surgery | 3 days after surgery
  Total number of PCEAs at 24, 48 and 72 hours after surgery
Rescue analgesic drug rates after 24, 48 and 72 hours after surgery | 3 days after surgery
  Rescue analgesic drug rates after 24, 48 and 72 hours after surgery
Adverse event( PONV, pruritus, hypotension ) rates at 24, 48 and 72 hours after surgery | 3 days after surgery
  Adverse event( PONV, pruritus, hypotension ) rates at 24, 48 and 72 hours after surgery
Local anaesthetic and opioid consumption | 3 days after surgery
  Local anaesthetic and opioid consumption
Patient satisfaction | 1 week after surgery
  Patient satisfaction score is from 0 to 100 points. The higher scores, the more satisfaction.
Length of hospital stay | 1 month after surgery
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Renchun Lai, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Renchun Lai, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bendixen M, Jorgensen OD, Kronborg C, Andersen C, Licht PB. Postoperative pain and quality of life after lobectomy via video-assisted thoracoscopic surgery or anterolateral thoracotomy for early stage lung cancer: a randomised controlled trial. Lancet Oncol. 2016 Jun;17(6):836-844. doi: 10.1016/S1470-2045(16)00173-X. Epub 2016 May 6. PMID 27160473
- [Result] Bertolaccini L, Fornaro G, Ciani O, Prisciandaro E, Crisci R, Tarricone R, Spaggiari L; VATS Group. The Impact of Surgical Experience in VATS Lobectomy on Conversion and Patient Quality of Life: Results from a Comprehensive National Video-Assisted Thoracic Surgical Database. Cancers (Basel). 2023 Jan 8;15(2):410. doi: 10.3390/cancers15020410. PMID 36672359
- [Result] Rauma V, Andersson S, Robinson EM, Rasanen JV, Sintonen H, Salo JA, Ilonen IK. Thoracotomy and VATS Surgery in Local Non-Small-Cell Lung Cancer: Differences in Long-Term Health-Related Quality Of Life. Clin Lung Cancer. 2019 Sep;20(5):378-383. doi: 10.1016/j.cllc.2019.05.010. Epub 2019 May 16. PMID 31202692
- [Result] Ng A, Swanevelder J. Pain relief after thoracotomy: is epidural analgesia the optimal technique? Br J Anaesth. 2007 Feb;98(2):159-62. doi: 10.1093/bja/ael360. No abstract available. PMID 17251209
- [Result] Yegin A, Erdogan A, Kayacan N, Karsli B. Early postoperative pain management after thoracic surgery; pre- and postoperative versus postoperative epidural analgesia: a randomised study. Eur J Cardiothorac Surg. 2003 Sep;24(3):420-4. doi: 10.1016/s1010-7940(03)00345-2. PMID 12965314
- [Result] Amr YM, Yousef AA, Alzeftawy AE, Messbah WI, Saber AM. Effect of preincisional epidural fentanyl and bupivacaine on postthoracotomy pain and pulmonary function. Ann Thorac Surg. 2010 Feb;89(2):381-5. doi: 10.1016/j.athoracsur.2009.10.060. PMID 20103303
- [Result] Bishop B, Pearce B, Willshire L, Kilpin M, Howard W, Weinberg L, Tan C. High Frequency, Low Background Rate Extrapleural Programmed Intermittent Bolus Ropivacaine Provides Superior Analgesia Compared with Continuous Infusion for Acute Pain Management Following Thoracic Surgery: A Retrospective Cohort Study. Anesth Pain Med. 2019 Oct 9;9(5):e97052. doi: 10.5812/aapm.97052. eCollection 2019 Oct. PMID 31903338
- [Result] Ueda K, Ueda W, Manabe M. A comparative study of sequential epidural bolus technique and continuous epidural infusion. Anesthesiology. 2005 Jul;103(1):126-9. doi: 10.1097/00000542-200507000-00019. PMID 15983464
- [Result] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Result] Hussain N, Lagnese CM, Hayes B, Kumar N, Weaver TE, Essandoh MK, Reno J, Small RH, Abdallah FW. Comparative analgesic efficacy and safety of intermittent local anaesthetic epidural bolus for labour: a systematic review and meta-analysis. Br J Anaesth. 2020 Oct;125(4):560-579. doi: 10.1016/j.bja.2020.05.060. Epub 2020 Jul 21. PMID 32703549
- [Result] Wydall S, Zolger D, Owolabi A, Nzekwu B, Onwochei D, Desai N. Comparison of different delivery modalities of epidural analgesia and intravenous analgesia in labour: a systematic review and network meta-analysis. Can J Anaesth. 2023 Mar;70(3):406-442. doi: 10.1007/s12630-022-02389-9. Epub 2023 Jan 31. PMID 36720838
- [Result] Capogna G, Camorcia M, Stirparo S, Farcomeni A. Programmed intermittent epidural bolus versus continuous epidural infusion for labor analgesia: the effects on maternal motor function and labor outcome. A randomized double-blind study in nulliparous women. Anesth Analg. 2011 Oct;113(4):826-31. doi: 10.1213/ANE.0b013e31822827b8. Epub 2011 Jul 25. PMID 21788309
- [Result] Leone Roberti Maggiore U, Silanos R, Carlevaro S, Gratarola A, Venturini PL, Ferrero S, Pelosi P. Programmed intermittent epidural bolus versus continuous epidural infusion for pain relief during termination of pregnancy: a prospective, double-blind, randomized trial. Int J Obstet Anesth. 2016 Feb;25:37-44. doi: 10.1016/j.ijoa.2015.08.014. Epub 2015 Oct 1. PMID 26431778
- [Result] Hogan Q. Distribution of solution in the epidural space: examination by cryomicrotome section. Reg Anesth Pain Med. 2002 Mar-Apr;27(2):150-6. doi: 10.1053/rapm.2002.29748. PMID 11915061
- [Result] Cole J, Hughey S. Bolus epidural infusion improves spread compared with continuous infusion in a cadaveric porcine spine model. Reg Anesth Pain Med. 2019 Sep 27:rapm-2019-100818. doi: 10.1136/rapm-2019-100818. Online ahead of print. PMID 31563882
- [Result] Lee SS, Baek JH, Park SJ, Kim HJ, Kim HY, Byeon GJ. Comparison of programmed intermittent epidural bolus injection and continuous epidural injection in controlling nighttime pain and improving sleep quality after thoracotomy. Medicine (Baltimore). 2022 Nov 11;101(45):e31684. doi: 10.1097/MD.0000000000031684. PMID 36397414
- [Result] Higashi M, Shigematsu K, Nakamori E, Sakurai S, Yamaura K. Efficacy of programmed intermittent bolus epidural analgesia in thoracic surgery: a randomized controlled trial. BMC Anesthesiol. 2019 Jun 15;19(1):107. doi: 10.1186/s12871-019-0780-0. PMID 31200641
- [Result] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Result] Myles PS, Myles DB. An Updated Minimal Clinically Important Difference for the QoR-15 Scale. Anesthesiology. 2021 Nov 1;135(5):934-935. doi: 10.1097/ALN.0000000000003977. No abstract available. PMID 34543410
- [Result] Finnerty DT, McMahon A, McNamara JR, Hartigan SD, Griffin M, Buggy DJ. Comparing erector spinae plane block with serratus anterior plane block for minimally invasive thoracic surgery: a randomised clinical trial. Br J Anaesth. 2020 Nov;125(5):802-810. doi: 10.1016/j.bja.2020.06.020. Epub 2020 Jul 11. PMID 32660716
- [Result] Moorthy A, Ni Eochagain A, Dempsey E, Wall V, Marsh H, Murphy T, Fitzmaurice GJ, Naughton RA, Buggy DJ. Postoperative recovery with continuous erector spinae plane block or video-assisted paravertebral block after minimally invasive thoracic surgery: a prospective, randomised controlled trial. Br J Anaesth. 2023 Jan;130(1):e137-e147. doi: 10.1016/j.bja.2022.07.051. Epub 2022 Sep 13. PMID 36109206